CLINICAL TRIAL: NCT02256878
Title: A Study to Evaluate the Effect of a Single Oral Dose and Multiple Oral Doses of 500 mg of BIRT 2584 XX Tablets on the Pharmacokinetic Parameters of Amitriptyline and Nortriptyline in Healthy Male and Female Subjects
Brief Title: Study to Evaluate the Effect Single and Multiple Oral Doses of BIRT 2584 XX Tablets on the Pharmacokinetic Parameters of Amitriptyline and Nortriptyline in Healthy Male and Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1206.12
Record Dates: First submitted 2014-10-02; First posted 2014-10-06 (Estimated); Last update posted 2014-10-06 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
MeSH Terms: interventions — Amitriptyline

ARMS (1):
- BIRT 2584 XX + Amitriptyline (Experimental): BIRT 2584 XX:
  Days 1 and 2: twice daily (bid) Days 3 to 21: once daily (qd)
  Amitriptyline:
  Single dose on day -8, day 1, and day 15
  Interventions: Drug: BIRT 2584 XX; Drug: Amitriptyline

INTERVENTIONS:
Drug: BIRT 2584 XX
Drug: Amitriptyline
  Other Names: Saroten®

SUMMARY:
The objective of the study was evaluate that there is no clinically relevant interaction between amitriptyline (or its metabolite nortriptyline) and BIRT 2584 XX (or its metabolite BI 610100) when BIRT 2584 XX is administered as a tablet formulation to near steady state in an estimated high therapeutic dose. Pharmacokinetics (PK) of amitriptyline and nortriptyline were measured before dosing of BIRT 2584 XX, after the first dose of BIRT 2584 XX, and after repeated doses of BIRT 2584 XX near steady state

ELIGIBILITY:
Inclusion Criteria:

* Healthy female or male volunteers as determined by the results of screening based upon a complete medical history, including physical examination, measurement of vital signs (Blood Pressure (BP), Pulse Rate (PR)), 12-lead ECG, and clinical laboratory tests
* Age ≥ 18 and ≤ 55 years
* BMI ≥ 18.5 and ≤ 29.9 kg/m2 (body mass index)
* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and the local legislation

Exclusion Criteria:

* Any finding of the medical examination (including BP, PR, and ECG) deviating from normal and of clinical relevance
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunologic, hematologic, oncologic or hormonal disorders
* Surgery of gastrointestinal tract (except appendectomy)
* Diseases of the Central Nervous System (CNS) (such as epilepsy) or psychiatric disorders or neurological disorders
* Relevant history of orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Intake of drugs with a long half-life (> 24 h) within 1 month prior to administration of the study drug or during the trial
* Use of any drugs which might influence the results of the trial within 10 days prior to study drug administration or expected during the trial
* Participation in another trial with an investigational drug within 2 months prior to administration or expected during the trial
* Smoker (>10 cigarettes or >3 cigars or >3 pipes/day); inability to abstain from smoking within 5 days before first drug administration until completion of the trial
* Alcohol abuse (>60 g/day)
* Drug abuse
* Blood donation or loss >400 mL, within 1 month prior to study drug administration or expected during the trial
* Clinically relevant laboratory abnormalities

For male subjects:

* Male subjects whose sexual partners are currently not using an adequate method of contraception that would prospectively be maintained during the study, are to be excluded
* Male subjects who are not willing to use condoms are to be excluded

For female subjects:

* Pregnancy
* Positive pregnancy test
* No highly safe method of contraception in women of childbearing potential (in this context, only sterilization or male partner sterilization is considered a highly safe method of contraception). Hormonal contraceptives are not considered adequate due to possible drug interaction with BIRT 2584 XX
* Lactation period

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2004-08; Primary Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
AUC0-∞ of amitriptyline (area under the concentration-time curve of amitriptyline in plasma over the time interval from 0 extrapolated to infinity) | up to 15 days
AUC0-∞ ratio of amitriptyline/nortriptyline | up to 15 days

SECONDARY OUTCOMES:
AUC0-∞ of amitriptyline (area under the concentration-time curve of amitriptyline in plasma over the time interval from 0 extrapolated to infinity) | Day 1
  1 hour after BIRT 2584 XX
Cmax of amitriptyline (maximum concentration of amitriptyline in plasma) | up to 15 days
AUC0-∞ of nortriptyline (area under the concentration-time curve of nortriptyline in plasma over the time interval from 0 extrapolated to infinity) | up to 15 days
Cmax of nortriptyline (maximum concentration of nortriptyline in plasma) | up to 15 days
AUC0-∞ ratio of amitriptyline/nortriptyline | Day 1
  1 hour after BIRT 2584 XX
AUC0-tz (area under the concentration-time curve of the analytes in plasma over the time interval from 0 to the time of the last quantifiable data point) | up to 15 days
tmax (time from dosing to the maximum concentration of the analytes in plasma) | up to 15 days
λz (terminal rate constant of the analytes in plasma) | up to 15 days
t1/2 (terminal half-life of the analytes in plasma) | up to 15 days
MRTpo (mean residence time of the analytes in the body after po administration) | up to 15 days
CL/F (apparent clearance of the analytes in the plasma after extravascular administration) | up to 15 days
Vz/F (apparent volume of distribution during the terminal phase following an extravascular dose) | up to 15 days
Pre-dose levels of BIRT 2584 XX and BI 610100 | up to 15 days
Number of subjects with adverse events | up to 57 days
Number of subjects with abnormal changes in laboratory parameters | up to 28 days
Assessment of tolerability by investigator on a 4-point scale | Day 28